CLINICAL TRIAL: NCT02211482
Title: Dolutegravir-Lamivudine as Dual Therapy in Naive HIV-Infected Patients: A Pilot Study
Acronym: PADDLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Pedro Cahn, PhD, Fundación Huésped
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-18
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infected patients; dual therapy
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dolutegravir , lamivudine (Other): Dolutegravir 50 mg QD plus lamivudine 300 mg QD
  Interventions: Drug: dolutegravir, lamivudine

INTERVENTIONS:
Drug: dolutegravir, lamivudine — single arm
  Other Names: dolutegravir; lamivudine

SUMMARY:
The purpose of this study is to evaluate the antiviral efficacy, safety and tolerability of dual therapy with 3TC and DTG as initial therapy among naïve HIV patients

DETAILED DESCRIPTION:
The purpose of this study is to compare the antiviral efficacy, safety and tolerability of dual therapy with 3TC and DTG as initial therapy among naïve HIV patients.

Data collected in this study would inform the development of larger studies designed to evaluate metabolic and long term safety, impact on inflammatory biomarkers, efficacy, safety and cost effectiveness of this strategy among naïve and suppressed patients.

Primary endpoint:Proportion of patients with HIV-1 RNA levels of less than 50 copies/mL at week 48.

Secondary endpoints: Frequency, type and severity of adverse events and laboratory abnormalities, Proportion of patients with HIV-1 RNA <1000 copies/mL at week 12, Proportion of patients with HIV-RNA <400 at week 24 Number and type of resistance mutations in case of virologic failure (defined as a confirmed viral above 400 copies/mL after week 24 copies/mL or viral rebound at any timepoint) Changes in CD4+ lymphocyte count between baseline and 48 weeks, Estimation of the viral decay compared to historical data.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Documented HIV-1 infection (positive ELISA plus a confirmatory Western Blot; or plasma HIV-1 RNA ≥10,000 copies/mL)
3. Voluntarily signed and dated , IRB / IEC approved informed consent form
4. Agrees not to take any other medication during the study
5. Screening HIV RNA >5,000 copies/mL and ≤ 100,000 copies/ml
6. Naïve to ARV therapies
7. CD4 ≥200 cells/mL
8. Subjects can comply with protocol requirements
9. Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the trial
10. Patient is a male or a female not breastfeeding or pregnant
11. A female, may be eligible if she:

    1. is of non-child-bearing potential
    2. is of child-bearing potential with a negative pregnancy test at Screening and Day 1 and agrees to use one of the following methods:

       * Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after
       * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
       * IUD and male condom
       * Male partner sterilization confirmed and male condom
       * Approved hormonal contraception and male condom
       * Any other method with published data showing that the expected failure rate is <1% per year and use male condom
       * Any contraception method must be used for at least 2 weeks after discontinuation of IP

Exclusion Criteria:

1. Genotypic resistance to lamivudine at screening,as per IAS -USA Panel 2013 2. Alcohol or drug use that might impact on adherence 3. Subjects positive for Hepatitis B at screening (+HBsAg), or anticipated need for Hepatitis C virus (HCV) therapy during the study 4. Lactating, pregnancy or fertile women willing to be pregnant 5. Concomitant use of lowering lipid drugs, interferon, interleukin-2, cytotoxic chemotherapy, Dofetilide (or pilsicainide ) or immunosuppressors at study entry 6. Grade 4 lab abnormalities 7. Primary HIV infection (indeterminate WB or previous negative HIV in the last 6 months.) 8. Opportunistic infection (CDC C category) or other disease and/or clinical condition that, in the investigator's opinion, would compromise the patient's safety or outcome of the study; including malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia 9. Subjects who in the investigator's judgment, poses a significant suicidality risk 10. History or presence of allergy to the study drugs or their components or drugs of their class 11. Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses or treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening or exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product 12. Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound 13. Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN), or ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin) 14. Creatinine clearance of <50 mL/min via Cockcroft-Gault method 15. Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Efficacy Outcome Measure | 48 weeks
  Percentage of Participants with HIV-1 RNA levels of less than 50 copies/mL at week 48 by ITT analysis

SECONDARY OUTCOMES:
safety | 48 week
  Frequency, type and severity of adverse events and laboratory abnormalities

OTHER OUTCOMES:
efficacy | 24 weeks
  Proportion of patients with HIV-RNA <400 at week 24
safety | 48 weeks
  change in lipid profile between baseline and week 48.
efficacy | 12 weeks
  Proportion of patients with HIV-1 RNA <1000 copies/mL at week 12
Number and type of resistance mutations in case of virologic failure (defined as a confirmed viral above 400 copies/mL after week 24 copies/mL or viral rebound at any timepoint) | 48 weeks
  Number and type of resistance mutations in case of virologic failure (defined as a confirmed viral above 400 copies/mL after week 24 copies/mL or viral rebound at any timepoint)
efficacy | 48 weeks
  Changes in CD4+ lymphocyte count between baseline and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cahn, PhD, Principal Investigator — Fundacion Huesped
Locations (1):
- Fundacion Huesped, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
to publish week 48 study results

REFERENCES:
- [Derived] Cahn P, Rolon MJ, Figueroa MI, Gun A, Patterson P, Sued O. Dolutegravir-lamivudine as initial therapy in HIV-1 infected, ARV-naive patients, 48-week results of the PADDLE (Pilot Antiretroviral Design with Dolutegravir LamivudinE) study. J Int AIDS Soc. 2017 May 9;20(1):21678. doi: 10.7448/IAS.20.01.21678. PMID 28537061